CLINICAL TRIAL: NCT07273422
Title: Evaluation of Self-powered Smart Insoles
Brief Title: Novel Self-charging, Medical-Grade Smart Insoles With AI/ML Edge Computing to Monitor Biometrics.
Status: Recruiting | Type: Observational
Sponsor: Spectrum Ergonomics and Occupational Health Services (Industry)
Collaborators: University of Utah (Other); United States Air Force Research Laboratory (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB_00176473; SEMI NBMC, NB18-24-44 (Other Grant/Funding Number: USAFRL)
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: No Applicable Condition; Study of Physiologic Monitor Alarms
Keywords: remote patient monitoring, energy harvesting,

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Males and female ages 18-100 years old and ambulatory
  Interventions: Other: Observational with data collected

INTERVENTIONS:
Other: Observational with data collected — Observational with data collection from sensors in insole

SUMMARY:
This study will evaluate the effectiveness of newly developed self-powered, smart insoles that will be used for remote patient monitoring (RPM) for both military and civilian populations. The present study is part of a project funded by SEMI and the Air Force Research Laboratory (AFRL).

DETAILED DESCRIPTION:
The present study, funded jointly by SEMI and the AFRL, is intended to evaluate the comfort, durability, and sensor accuracy of the smart insoles and associated mobile app. The study will evaluate both generation 1.0 and generation 2.0 of the smart insole. The primary difference between the two generations is the that gen 2.0 will use an improved energy harvester for power generation.

The present study is structured in two phases. Phase 1 will evaluate gen 1.0 of the insole in a pilot study at the University of Utah (U of U) with 10 subjects. The subjects will be asked to wear the insole while walking at different speeds on an instrumented treadmill in the Motion Core Analysis Facility at the University of Utah and asked to walk over a ½ mile course on the U of U campus. This study will be overseen by Dr. Shad Roundy.

Phase 2 will evaluate gen 2.0 of the insole. A pilot study will take place at the U of U and will mimic the phase 1 study with 10 subjects. Again, the study will be overseen by Dr. Shad Roundy. This will be followed up by a larger field study with 100 subjects who will be asked to take the insoles home and wear them over the course of 4 weeks. The field study will be overseen by Dr. Jeff Hiserman at Spectrum Ergonomics.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is generally health and between 18 and 90 year of age at time of signing consent.
2. Participant must be available for 4 visits to Spectrum Ergonomics over a 4-week period, one visit per week.

   -

Exclusion Criteria:

* Age of Participants: 18-90

Sample Size:

At Utah:

All Centers: 120

Inclusion Criteria:

Inclusion criteria for Phase 1 and Phase 2 pilot studies at UofU

1. Participant is generally healthy and between 18 and 90 years of age at time of signing consent 2. Participant must be able to walk comfortably for 1 mile. 3. Will seek 5 male and 5 female participants. Inclusion criteria for Phase 2 field studies conducted by Spectrum Ergonomics

1. Participant is generally health and between 18 and 90 year of age at time of signing consent.
2. Participant must be available for 4 visits to Spectrum Ergonomics over a 4-week period, one visit per week.

Exclusion Criteria:

Exclusion Criteria for Phase 1 and Phase 2 pilot studies at UofU

* Flat feet (Pes planus)
* Unilateral leg amputee
* Females who are pregnant, < 3 months postpartum, or currently lactating.
* Major surgery < 6 months or minor surgery < 3 months before enrollment.
* Major infections such as sepsis or pneumonia < 3 months before enrollment.
* Myocardial infarction or heart failure < 5 years or less before enrollment.
* Ankle fusion or total replacement
* Morbid obesity BMI > 40.

Exclusion Criteria for Phase 2 field study at Spectrum Ergonomics

* Flat feet (Pes planus) or high arches (Pes cavus)
* Unilateral leg amputee.
* Brittle Diabetes- hard-to-control diabetes (also called labile diabetes), which is characterized by wide variations in blood glucose in which blood glucose levels can quickly move from too high (hyperglycemia) to too low (hypoglycemia).
* Peripheral neuropathy.
* Loss of sensation in the sole of foot.
* Open wound on the foot.
* Females who are pregnant, < 3 months postpartum, or currently lactating.
* Ankle fusion or total replacement
* Major surgery < 6 months or minor surgery < 3 months before enrollment.
* Major infections such as sepsis or pneumonia < 3 months before enrollment.
* Myocardial infarction or heart failure < 1 years before enrollment.
* Morbid obesity BMI > 40.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the clinic's patient population, their family and friends, and from the general public in the northcentral Pennsylvania region.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The present study is intended to evaluate the safety of the sensors embedded in the smart insoles and their accuracy in measuring biomarkers. | "From enrollment to the end of observations at 4 weeks"
  The sensors will measure: Pulse Oxygen as the percentage saturation of oxygen carried in the red blood cells.

SECONDARY OUTCOMES:
The present study is intended to evaluate the safety of the sensors embedded in the smart insoles and their accuracy in measuring biomarkers. | Time Frame: "From enrollment to the end of observations at 4 weeks"
  Description: The sensors will measure: Heart Rate and Heart Rate Variability in beats per minute.

OTHER OUTCOMES:
The present study is intended to evaluate the safety of the sensors embedded in the smart insoles and their accuracy in measuring biomarkers. | Time Frame: "From enrollment to the end of observations at 4 weeks"
  Description: The sensors will measure: Body temperature as measured in degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Andosca, PhD, Principal Investigator — Inviza Health
Locations (1):
- Spectrum Ergonomics and Occupational Health Services, Williamsport, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The data will be shared as group data, divided into various groups, i.e. age and gender.